CLINICAL TRIAL: NCT02236429
Title: Vaginal Flora Transplantation for Recurrent Bacterial Vaginosis
Brief Title: Vaginal Flora for Treatment of Bacterial Vaginosis
Acronym: VFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VFT-HMO-CTIL
Record Dates: First submitted 2014-09-07; First posted 2014-09-10 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Bacterial Vaginitis
Keywords: bacterial vaginitis; vaginal flora; microbiome
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recurrent bacterial vaginitis (Experimental)
  Interventions: Biological: vaginal flora transplant

INTERVENTIONS:
Biological: vaginal flora transplant

SUMMARY:
Bacterial vaginosis (BV) is the most common vaginal infection in women. It is caused by a vaginal bacterial imbalance. Treatment with antibiotics is the standard of care but there is a high rate of recurrence. Almost half of women successfully treated suffer a recurrence within three months. Complications include risk factors for premature birth, increased transmission of sexually transmitted diseases and higher risk for carcinoma of cervix. The investigators proposed study is a cost effective treatment based on returning the normal microbial balance to the vagina. The investigators propose to transfer normal vaginal flora from healthy individuals to women with BV and thus restore normal vaginal flora and cure this disorder.

ELIGIBILITY:
Inclusion Criteria:

* recurrent BV (4 or more incidences in the past year)
* recurrence of BV in less than 2 months of antibiotic treatment or need for prophylactic antibiotic
* 3/4 Amsel criteria and Nugent criteria greater or equal to 7

Exclusion Criteria:

* pregnancy or planned pregnancy during the study period
* other known diseases
* carriers of Hep B and C
* HIV or syphilis positive

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
relief of bacterial vaginosis | 12 month
  Clinical cure, i.e., absence of vaginal discharge and malodor

SECONDARY OUTCOMES:
Laboratory parameters | 12 months
  absence of all Amsel criteria and Nugent score<3.

CONTACTS AND LOCATIONS:
Overall Officials: Ahinoam Lev-Sagie, MD, Principal Investigator — Hadassah Mediocal Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lev-Sagie A, Goldman-Wohl D, Cohen Y, Dori-Bachash M, Leshem A, Mor U, Strahilevitz J, Moses AE, Shapiro H, Yagel S, Elinav E. Vaginal microbiome transplantation in women with intractable bacterial vaginosis. Nat Med. 2019 Oct;25(10):1500-1504. doi: 10.1038/s41591-019-0600-6. Epub 2019 Oct 7. PMID 31591599